CLINICAL TRIAL: NCT02684136
Title: A Double-blind, Crossover, Study to Compare the Hypnotic, Daytime Sleepiness/Fatigue, and Pain Effects of Nighttime Administration of Suvorexant 20 mg Versus Placebo in Patients With Fibromyalgia and Comorbid Insomnia
Brief Title: Suvorexant in Insomnia Co-morbid With Fibromyalgia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: reduced ability to recruit sufficient number of patients
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Timothy Roehrs, PhD, Senior Bioscientist, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FM16
Record Dates: First submitted 2016-01-22; First posted 2016-02-17 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-04

CONDITIONS: Insomnia; Fibromyalgia
Keywords: insomnia; fibromyalgia; polysomnography; pain management
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fibromyalgia; Agnosia | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- suvorexant (Experimental): 9 nights of 20 mg suvorexant
  Interventions: Drug: suvorexant
- placebo (Placebo Comparator): 9 nights placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: suvorexant — suvorexant 20 mg taken before sleep
  Other Names: belsomra
  Arms: suvorexant
Drug: placebo — placebo taken before sleep
  Other Names: matching placebo
  Arms: placebo

SUMMARY:
This study will compare sleep, pain and daytime sleepiness/fatigue in people with insomnia co-morbid with fibromyalgia while treated short-term with suvorexant 20 mg versus placebo.

DETAILED DESCRIPTION:
It has now become clear that the relation of sleep and pain is bidirectional; acute and chronic pain is associated with disturbed sleep and disturbed sleep enhances pain. Experimental studies have shown that reduced and fragmented sleep in pain-free normals increases their pain sensitivity and daily self-report studies in chronic pain patients have shown a poor night of sleep is followed by enhanced next-day pain. In mediation analyses of large clinical data sets it is found that the sleep-pain side of the bidirectional relation, as opposed to the pain-sleep side, accounts for the greater variance. These data then would suggest that improving sleep in chronic pain disorders should attenuate daytime pain.

Most of the drugs used to treat chronic pain facilitate inhibitory central nervous system mechanisms as their primary mechanism of action. Suvorexant, recently approved by the FDA for the treatment of insomnia characterized by difficulties with sleep onset and sleep maintenance, has a unique mechanism of action. Suvorexant is a selective antagonist for orexin receptors (OX1R and OX2R). Orexins are considered to be involved in arousal and maintenance of the waking state.

As such, suvorexant may provide unique clinical benefit as a treatment in chronic pain conditions with co-morbid insomnia, and specifically for fibromyalgia with its putative central hyperarousal and hypersensitization. Thus, this project proposes to study objective and clinical measures of sleep, pain, and daytime sleepiness and fatigue in patients with fibromyalgia and co-morbid insomnia while treated short-term with suvorexant 20 mg versus placebo.

Those qualifying will receive suvorexant 20 mg and placebo for each of 9 nights in a cross over design with 7 nights of washout between treatments. Overnight sleep recordings (PSGs) will be collected on nights 7 and 8 of each crossover treatment arm to determine objective sleep measures. During the day following night 7 in each arm, a Multiple Sleep Latency Test (MSLT) at 1000, 1200, 1400, and 1600 hr will be conducted and nociceptive sensitivity [finger withdrawal latency (FWL)] testing to a radiant heat stimulus (1100 and 1500 hr) will be conducted on day 1 and day 8. Self-reported mood and pain indices will also be completed prior to each FWL test.

Primary outcomes to be measured include PSG sleep efficacy and FWL response on both conditions (suvorexant 20 mg versus placebo).

ELIGIBILITY:
Inclusion Criteria:

* meet Diagnostic and Statistical Manual 5th ed criteria for insomnia
* meet American College of Rheumatology criteria for fibromyalgia
* otherwise good psychiatric and stable physical health

Exclusion Criteria:

* other primary sleep disorders
* pain symptoms unrelated to fibromyalgia
* current pregnancy or breast-feeding

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-01; Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Roehrs, PhD, Principal Investigator — Henry Ford Health System; Thomas Roth, PhD, Study Chair — Henry Ford Health System
Locations (1):
- HFHS Sleep Disorders Ctr, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Roehrs T, Diederichs C, Gillis M, Burger AJ, Stout RA, Lumley MA, Roth T. Nocturnal sleep, daytime sleepiness and fatigue in fibromyalgia patients compared to rheumatoid arthritis patients and healthy controls: a preliminary study. Sleep Med. 2013 Jan;14(1):109-15. doi: 10.1016/j.sleep.2012.09.020. Epub 2012 Nov 11. PMID 23149217
- [Derived] Roehrs T, Withrow D, Koshorek G, Verkler J, Bazan L, Roth T. Sleep and pain in humans with fibromyalgia and comorbid insomnia: double-blind, crossover study of suvorexant 20 mg versus placebo. J Clin Sleep Med. 2020 Mar 15;16(3):415-421. doi: 10.5664/jcsm.8220. Epub 2020 Jan 14. PMID 31992394

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant First, Then Placebo: 9 nights of 20 mg suvorexant first, then 9 nights of placebo suvorexant: suvorexant 20 mg taken before sleep; placebo taken before sleep
- Placebo First, Then Suvorexant: 9 nights placebo first, washout, then 9 nights of 20 mg suvorexant: suvorexant 20 mg taken before sleep; placebo taken before sleep
Period: First Intervention (9 Nights)
Arm/Group | Suvorexant First, Then Placebo | Placebo First, Then Suvorexant
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Suvorexant First, Then Placebo | Placebo First, Then Suvorexant
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (9 Nights)
Arm/Group | Suvorexant First, Then Placebo | Placebo First, Then Suvorexant
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: this is a crossover study
Groups:
- All Study Participants: this is a crossover study with 20 mg suvorexant and placebo each administered for 9 nights
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Total Sleep Time [Mean (Standard Deviation); unit: min of total sleep time on a 8-hr PSG] — minutes of total sleep time on a 8-hr PSG
  min of total sleep time on a 8-hr PSG | 346.9 (52.32)

OUTCOME MEASURES:

1. Primary Outcome: Polysomnographic Assessment of Sleep
Description: total sleep time on 8 hr standard sleep recording
Time Frame: continuous sleep recording from 11pm to 7am on night 8
Population: this is crossover study so all 10 Ss received both placebo and suvorexant
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
min | 429.3 (29.4) | 400.5 (57.3)
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p < 0.05, ANCOVA; baseline used as covariate

2. Secondary Outcome: Daytime Pain Sensitivity
Description: finger withdrawal response to a radiant heat stimulus when pain is first experienced
Time Frame: mean of tests at 1100 and 1500 hrs on both day 1 and day 8
Population: this is a crossover study so all 10 Ss received placebo and suvorexant
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 10 | 10
sec | 15.8 (5.4) | 14.7 (4.9)
Statistical Analysis 1: Comparison: Suvorexant vs Placebo; Test type: Superiority; p < 0.05, ANCOVA — baseline used as covariate

ADVERSE EVENTS:
Time Frame: nightly over the 9 nights
Description: this is a crossover study and all 10 Ss were at risk in the placebo and suvorexant arms
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=10) | Placebo (N=10)
headache (Nervous system disorders) | 8 (17) | 3 (3) — headache, dizziness, residual sedation - adverse event terms can not be separated

LIMITATIONS AND CAVEATS:
Study closed after 18 moinths due to difficulty recruiting additional subjects beyond the 10 completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT02684136/Prot_SAP_000.pdf